CLINICAL TRIAL: NCT06481163
Title: A Phase 2 Multicentre, Open-label Study to Evaluate the Efficacy, Safety and Tolerability, and Pharmacokinetics of 14 -28 Days Telacebec Treatment in Adult Participants With Buruli Ulcer.
Brief Title: Telacebec (T) Treatment in Adults With Buruli Ulcer (BU).
Acronym: Treat BU
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Barwon Health (Other Government)
Collaborators: Global Alliance for TB Drug Development (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TBA-BU-01
Record Dates: First submitted 2024-06-21; First posted 2024-07-01 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-11

CONDITIONS: Buruli Ulcer
Keywords: lesion; ulcer; Buruli Ulcer; telacebec; Q203
MeSH Terms: conditions — Buruli Ulcer; Ulcer | interventions — telacebec

STUDY DESIGN:
Intervention Model Description: Open Label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- 300 mg Telacebec per day (Experimental): Telacebec will be administered orally with food or within 30 minutes after food once daily for 14-28 consecutive days.
  Interventions: Drug: Telacebec

INTERVENTIONS:
Drug: Telacebec — The test product will be supplied as Telacebec 100mg tablets.
  Other Names: Q203

SUMMARY:
The goal of this interventional clinical trial is to determine if treatment with 2-4 weeks of telacebac (T) will completely heal lesions in participants with Buruli ulcer (BU) by 52 weeks after treatment initiation, without relapse and/or surgery. Males and females age 18 and older will be included.

• Participants will attend visits every 2 weeks during treatment and thereafter every 2 weeks until week 24 Thereafter they will be followed by visits at weeks 30, 40, and 52. From week 10 to week 52, if the lesion has healed, follow-up visits may be remote.

DETAILED DESCRIPTION:
This is an open label single arm (telacebec), phase 2 multi-centre, clinical trial. Eligible participants with clinically diagnosed BU, confirmed by polymerase chain reaction (PCR) or culture presence of MU infection Participants who meet entry criteria and give consent will attend a baseline enrolment visit (Day 1), then visits every week for 2 weeks during treatment (weeks 2, and 4). Thereafter they will be followed up every 2 weeks until week 24, followed by visits at weeks 30, 40, and 52.

BU lesion management will be provided to all trial participants. In case of participant early withdrawal from the trial during or after the treatment period, participants will be treated per the investigational site and/or country BU treatment guidelines.

A Data Review Committee (DRC) will be established to review efficacy and safety data. Enrolment and enrolled participants will continue the study whilst the DRC reviews are ongoing.

ELIGIBILITY:
Major Inclusion Criteria:

* Clinical diagnosis of BU
* Positive PCR or culture for confirmation of presence of mycobacterium ulcerans (MU).

Major Exclusion Criteria:

* Participants with the following known or suspected medical conditions:

  1. Any non BU related condition where participation in the study, as judged by the Investigator, could compromise the well-being of the participant or prevent, limit or confound protocol specified treatment and assessments.
  2. History or current ascites, jaundice, myasthenia gravis, clinically significant renal dysfunction [estimated glomerular filtration rate (eGFR) < 30 mls/min],
  3. History of previous BU in the previous 12 months (except current infection)
* Planned/expected to require curative intent excision surgery, defined as excision of lesion which may include surrounding macroscopically healthy tissue with the aim of helping to sterilize the wound rather than improve wound healing alone, for their BU during the entire study period. Simple removal of necrotic slough and skin grafting is considered normal wound care and allowed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2024-07-09 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Rate of complete lesion healing by 52 weeks from treatment initiation. | 52 weeks from treatment initiation
  Ulcerated Lesions: Healing and re-epithelialisation of ulcerated area with stable scar formation. Non-ulcerated Lesions: resolution of induration of skin.
  Complete healing rate will be summarized as percentage with corresponding Clopper-Pearson 95% confidence interval.

SECONDARY OUTCOMES:
Median time to healing | 52 weeks from treatment initiation
  Kaplan-Meier methods will be applied to estimate median time to healing.
Recurrence rate within 52 weeks from treatment initiation | 52 weeks from treatment initiation
  Complete lesion healing followed by a recurrent lesion at the same site or a new lesion appearing at a separate site, detected within 52 weeks of treatment initiation, that is culture positive and not judged to be due to a paradoxical response to telacebec treatment on clinical and/or histological findings.
Treatment failure rate within 52 weeks from treatment initiation | 52 weeks from treatment initiation
  Lack of complete healing within the 52 weeks observation period; Recurrence, Use of alternative buruli ulcer (BU) treatment, BU curative intent surgery
Safety and Tolerability | Time of first dose to 28 days after last dose of telacebec.
  Incidence of Treatment Emergent Adverse Events (TEAEs)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel O'Brien, MD, Principal Investigator — Barwon Health
Locations (2):
- Australia (2):
  - Barwon Health, Geelong, Victoria
  - Royal Melbourne Hospital, Melbourne

IPD SHARING:
Plan to Share IPD: Yes
On request and subject to approval by the Sponsor.